CLINICAL TRIAL: NCT03533673
Title: A Phase 1 Study of the Safety of AAV2/8-LSPhGAA (ACTUS-101) in Late-onset Pompe Disease
Brief Title: AAV2/8-LSPhGAA (ACTUS-101) in Late-Onset Pompe Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AskBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACT-CS101
Record Dates: First submitted 2018-04-13; First posted 2018-05-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pompe Disease
Keywords: Gene Therapy
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): A one-time intravenous infusion of ACTUS-101 (dose level 1)
  Interventions: Biological: ACTUS-101
- Cohort 2 (Experimental): A one-time intravenous infusion of ACTUS-101 (dose level 2)
  Interventions: Biological: ACTUS-101
- Cohort 3 (Experimental): A one-time intravenous infusion of ACTUS-101 (dose level 3)
  Interventions: Biological: ACTUS-101

INTERVENTIONS:
Biological: ACTUS-101 — Adeno-associated virus serotype 8 carrying the human GAA gene under the control of the LSP promoter.

SUMMARY:
Open-label, ascending dose trial of ACTUS-101 administered intravenously.

DETAILED DESCRIPTION:
This study will be a prospective, open-label trial designed to objectively assess the safety and bioactivity of ACTUS-101 in subjects diagnosed with Pompe disease, which is caused by a defect in acid α-glucosidase (GAA) gene. ACTUS-101 is intended to enable expression of a functional copy of the GAA gene in subject's hepatocytes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pompe disease by blood or skin fibroblast GAA assay and two pathogenic variants in the GAA gene,
* Age: Greater than or equal to 18 years at enrollment.
* Subjects are capable of giving written informed consent.
* Able to walk at least 100 meters on the 6MWT (with assistive devices permitted).
* FVC within the range of 30% to less 90% (inclusive) of predicted in the upright position.
* Subjects with a confirmed diagnosis of LOPD who have been treated with ERT for at least 104 weeks (inclusive) immediately preceding screening and receiving a stable dose of ERT for the 52-week period immediately preceding dosing.

Exclusion Criteria:

* Invasive ventilation required or noninvasive ventilation required while awake and upright.
* FVC <20% of predicted (supine).
* Received any live vaccination 2 months prior to study Day 1.
* Pregnant or nursing mothers.
* Serology consistent with exposure to HIV, or serology consistent with active hepatitis A, B or C infection. Any active liver disease.
* Active infection based upon clinical symptoms.
* Having started respiratory muscle strength training in the last 6 months prior to study day 1 or having discontinued respiratory muscle strength training in the 6-month period preceding study day 1, or having started respiratory strength training greater than 6 months prior to study day 1 and unwilling to continue for the first year of study participation.
* Received an investigational drug or participated in another interventional study within 90 days prior to Study Day 1. Additionally, subjects cannot participate in any other interventional clinical trial throughout the first 78 weeks after receiving ACTUS-101.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of patient reported Treatment Emergent Adverse Events (TEAEs) (safety and tolerability) | 78 weeks
  The incidence of patient reported TEAEs will be measured according to protocol specifications.
Incidence of patient reported Serious Adverse Events (SAEs) (safety and tolerability) | 78 weeks
  The incidence of patient reported SAEs will be measured according to protocol specifications.
Number of Participants With Abnormal Laboratory Values | 78 weeks
  Laboratory assessments will be performed (CBC, Chemistry, urinalysis, serology, anti-GAA antibody, T-cell response, GAA activity) and compared to baseline values.

SECONDARY OUTCOMES:
Muscle GAA Bioactivity | 78 weeks
  Muscle GAA activity will be compared to baseline by muscle biopsy
Serum GAA Bioactivity | 78 weeks
  Serum GAA activity will be compared to baseline by blood screening
Glycogen content in muscle | 78 weeks
  Muscle glycogen level compared to baseline by muscle biopsy
Anti-rhGAA antibody formation | 78 weeks
  Anti-rhGAA antibodies monitored by ELISA
Muscle Status Testing - 6 minute walk test | 78 weeks
  The 6-minute walk test will be performed and results compared to baseline.
Muscle Status Testing - Gross Motor Function Measure | 78 weeks
  The gross motor function measure (GMFM88) will be performed and the results compared to baseline.
Muscle Status Testing - Quick Motor Function Test (QMFT) Measure | 78 weeks
  Measurement of functional motor abilities using the Quick Motor Function Test (QMFT) will be performed and the results compared with baseline.
Muscle Status Testing - Gait, Stairs, Gower, Chair | 78 weeks
  The Gait, Stairs, Gower, Chair (GSGC) test will be performed and results compared to baseline.
Pulmonary Function Testing | 78 weeks
  Pulmonary function (forced vital capacity, FVC in liters of air) measured by spirometer in comparison to baseline.
Muscle Status Testing - Timed up and Go (TUG) | 78 weeks
  Measurement of functional motor abilities using the Timed up and Go (TUG) test will be performed and the results compared with baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith EC, Hopkins S, Case LE, Xu M, Walters C, Dearmey S, Han SO, Spears TG, Chichester JA, Bossen EH, Hornik CP, Cohen JL, Bali D, Kishnani PS, Koeberl DD. Phase I study of liver depot gene therapy in late-onset Pompe disease. Mol Ther. 2023 Jul 5;31(7):1994-2004. doi: 10.1016/j.ymthe.2023.02.014. Epub 2023 Feb 18. PMID 36805083